CLINICAL TRIAL: NCT03195153
Title: Effect of Allopurinol on Mono and Co-administration With Statins on Platelets Reactivity on Diabetic Patiets Treated With Aspirin and Insulin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Polacco Marina, MD, principal investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY OF ROME
Record Dates: First submitted 2017-05-28; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus Type 2 Platelets Reactivity Statin
MeSH Terms: interventions — Atorvastatin; Allopurinol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- statin only (Experimental): 30 DAYS OF STATIN THERAPY ATORVASTATIN 80 MG)
  Interventions: Drug: Atorvastatin 80mg
- allopurinol only (Experimental): 30 DAYS OF ALLOPURINOL (300 MG)
  Interventions: Drug: ALLOPURINOL 300 MG
- statin and allopurinol (Experimental): 30 DAYS OF CO-ADMINISTRATION OF ATORVASTATIN AND ALLOPURINOL
  Interventions: Drug: Atorvastatin 80mg AND allopurinol 300 mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — 30 DAYS OF atorvastatin 80 mg
  Arms: statin only
Drug: ALLOPURINOL 300 MG — 30 DAYS OF ALLOPURINOL 300 MG
  Arms: allopurinol only
Drug: Atorvastatin 80mg AND allopurinol 300 mg — 30 days of atorvastatin and allopurinol 300 mg
  Arms: statin and allopurinol

SUMMARY:
Diabetes mellitus is associated with an increased risk of cardiovascular disease. Substantial clinical and experimental evidence suggest that both diabetes and insulin resistance cause a combination of endothelial dysfunctions, which may diminish the anti-atherogenic role of the vascular endothelium. Therefore, in patients with diabetes or insulin resistance, endothelial dysfunction may be a critical early target for preventing atherosclerosis and cardiovascular disease. It has been implicated as an independent risk factor for cardiovascular disease and premature cardiovascular mortality for patients with type 1 and type 2 diabetes mellitus, as well as for patients with essential hypertension. A complete biochemical understanding of the mechanisms by which hyperglycemia causes vascular functional and structural changes associated with the diabetic milieu still eludes us. In recent years, the numerous biochemical and metabolic pathways postulated to have a causal role in the pathogenesis of diabetic vascular disease have been distilled into several unifying hypotheses. The role of chronic hyperglycemia in the development of diabetic microvascular complications and in neuropathy has been clearly established. However, the biochemical or cellular links between elevated blood glucose levels, and the vascular lesions remain incompletely understood. A number of trials have demonstrated that statins therapy as well as angiotensin converting enzyme inhibitors is associated with improvements in endothelial function in diabetes. Although antioxidants provide short-term improvement of endothelial function in humans, all studies of the effectiveness of preventive antioxidant therapy have been disappointing. Actually, control of hyperglycemia thus remains the best way to improve endothelial function and to prevent atherosclerosis and other cardiovascular complications of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patient;
* therapy with aspirin and insulin;
* patient well responders

Exclusion Criteria:

* not diabetic patient;
* patients in dual antiplatelet therapy;
* patient with severe renal failure;
* patient poor responders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-06-23 (Estimated); Study Completion 2017-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California] After 30 days of treatment with each drug | fter 30 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California]

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Rome, Roma, Italy